CLINICAL TRIAL: NCT02691130
Title: A Multicenter, Randomized, Double-blind, Active-controlled Phase 2b Trial [Part of EU-funded UNISEC Project] to Assess the Immunogenicity & Safety of a BiondVax's Influenza Vaccine (M-001) Followed by H5N1 Vaccine in Healthy Adults
Brief Title: Assess the Safety and Immunogenicity of M-001 as A Standalone Influenza Vaccine and as A H5N1 Vaccine Primer in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BiondVax Pharmaceuticals ltd. (Industry)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BVX-007
Record Dates: First submitted 2016-02-11; First posted 2016-02-25 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Influenza; Healthy
Keywords: influenza; vaccine; universal; peptide; prime; boost; HAI; CMI; UNISEC
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: M-001 0.5mg & H5N1 influenza vaccine (Experimental): Biological/Vaccine: Two Multimeric-001 administrations followed by H5N1 influenza vaccine
  Two administrations of non adjuvanted M-001, 0.5mg followed by 3mcg Alum/H5N1 influenza vaccine at intervals of 19-23 days
  Interventions: Biological: Multimeric 001 (M-001); Biological: H5N1 influenza vaccine
- B: M-001 1.0mg & H5N1 influenza vaccine (Experimental): Biological/Vaccine: Two Multimeric-001 administrations followed by H5N1 influenza vaccine
  Two administrations of non adjuvanted M-001, 1.0mg followed by 3mcg Alum/H5N1 influenza vaccine at intervals of 19-23 days
  Interventions: Biological: Multimeric 001 (M-001); Biological: H5N1 influenza vaccine
- C: Saline & H5N1 influenza vaccine (Placebo Comparator): Biological/Vaccine: Two saline administrations followed by H5N1 influenza vaccine
  Two administrations of saline followed by 3mcg Alum/H5N1 influenza vaccinated intervals of 19-23 days
  Interventions: Biological: H5N1 influenza vaccine; Biological: Saline

INTERVENTIONS:
Biological: Multimeric 001 (M-001) — Multimeric 001 is a recombinant protein comprising 9 conserved peptides from influenza A and B
  Arms: A: M-001 0.5mg & H5N1 influenza vaccine; B: M-001 1.0mg & H5N1 influenza vaccine
Biological: H5N1 influenza vaccine — Alum adjuvanted whole virion inactivated H5N1 vaccine produced by FluArt (Hungary)
Biological: Saline — 0.9% NaCl in double distilled water
  Arms: C: Saline & H5N1 influenza vaccine

SUMMARY:
"Multimeric-001" (M-001) contains conserved, common linear influenza epitopes that activate both cellular and humoral arms of the immune system against a wide variety of influenza A and B strains. Apart from its direct action, M-001 is an attractive candidate for priming immune responses to pandemic influenza vaccine in the adult population. The current clinical study was designed to assess M-001's standalone and priming action in subjects aged 18-60 years old.

This is a Phase IIb study comprising 222 participants. Eligible subjects were randomized to receive two sequential intramuscular injection of 0.5mg or 1.0mg M-001 (treatment), or two placebo (saline) injection, before receiving the sub optimal dose of H5N1 pandemic vaccine.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blind active-controlled Phase 2b study. 222 subjects will be randomized 1:1:1 into three groups to receive two sequential non-adjuvanted 0.5 mg or 1.0mg intramuscular injection of M-001 (treatment), or two placebo (saline) injection, before receiving the Alum adjuvanted H5N1 vaccine at a sub optimal dose of 3mcg. Hemagglutinin inhibition (HAI) will be evaluated at baseline and 3 weeks after H5N1 whole virion inactivated pandemic influenza vaccination as a measure of M-001's ability to enhance the humoral response. Cell mediated immune (CMI) responses will also be evaluated at baseline and after immunization with M-001 as a measure of M-001's standalone immunogenicity. The subjects will monitored for safety throughout the study until day 180.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 60 years, inclusive;
* Women of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to one year) and men must agree to practice adequate contraception (a combination of barrier plus hormone methods or intra uterine device (IUD) for women and a condom for men) throughout the study treatment and for at least up to day 51 (for female) and day 111 (for male) of the trial (i.e. 30 (for female) and 90 (for male) days after the last dose of the IMP);
* Is in good health, as determined by vital signs (heart rate, blood pressure, armpit temperature), blood chemistry test (electrolytes, renal/kidney function, liver function, C-reactive protein, complete blood count), medical history, general physical examination, self-reported illness and clinical judgment of the investigator;
* Able to understand and comply with planned study procedures;
* Provides signed informed consent form after receiving a detailed explanation of the study protocol prior to any study procedures.

Exclusion Criteria

A potential subject who meets any if the following criteria will be excluded from participation in this study:

* Has a known allergy to components of the vaccine (e.g. egg products).
* Has a history of severe reactions following immunization.
* Persons with immune deficiency/disorder, whether due to genetic defect, immunodeficiency disease, or immunosuppressive therapy.
* Has a positive urine pregnancy test prior to vaccination or women who are breastfeeding.
* Has a history of any of the following (reported by subjects):

  * Acute disseminated encephalomyelitis (ADEM);
  * Active neoplastic disease;
  * Asthma or severe allergic disease;
  * Bleeding disorders
  * Chronic Hepatitis B and/or C infection;
  * Chronic liver disease;
  * Diabetes mellitus;
  * Guillain-Barré syndrome;
  * HIV;
  * Rheumatoid arthritis or other autoimmune diseases;
  * Severe renal disease;
  * Transplant recipients;
  * Unstable or progressive neurological disorders.
* Receipt of medicines/treatments that may affect evaluation of immunogenicity such as:

  * Oral or parenteral steroids, high-dose inhaled steroids (greater than 800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs;
  * Immunoglobulin or other blood products (within the 3 months prior to vaccination in this study);
  * Experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study, or expects to receive an experimental agent (during the study period).
  * Influenza antiviral medication (within the 4 weeks prior to vaccination in this study).
* Has received any influenza vaccine within 6 months prior to vaccination in this study.
* Has influenza-like illness within 6 months prior to vaccination in this study.
* Has an acute illness, including an armpit temperature greater than 38 degrees Celsius (oC), within 1 week of vaccination.
* Has a history of alcohol or drug abuse.
* Any abnormal haematology values and/or serum chemistries judged by the Investigator as clinically significant.
* Ineligible subject based on the judgement of the investigator.
* In case there is uncertainty about the participant's medical status regarding any of the exclusion criteria mentioned, the participant's primary care physician will be consulted. Consultation of the primary care physician will only take place after having received written approval from the participant, and will concern medical information about exclusion criteria only.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
For each vaccine group the incidence rate of subjects with solicited AE(s) with 95% confidence interval | Day 0 to Day 42 (21 days after the last M-001 dosing)
  All subjects
For each vaccine group the percentage of subjects with SAE(s) with 95% confidence interval | Day 0 to Day 180 (study conclusion)
  All subjects
For each vaccine group the influenza-specific cellular immune responses evaluated by multi-parametric FACS analysis | Days 0 and 42 (21 days after the last M-001 dosing)
  All subjects

SECONDARY OUTCOMES:
For each vaccine group the antibody responses to the H5 vaccine strain evaluated by hemaglutination inhibition (HI) assay | Days 0 and 63 (21 days after the H5N1 immunization)
  All subjects

OTHER OUTCOMES:
Exploratory: For each vaccine group the antibody responses to the non-H5 vaccine strains evaluated by hemaglutination inhibition (HI) assay | Days 0 and 63 (21 days after the H5N1 immunization)
  All subjects
Exploratory: For each vaccine group the influenza-specific cellular immune responses evaluated by quantitative reserve transcription polymerase chain reaction (qRT-PCR) assay | Days 0, 42 and 63
  In all groups, in a subset of 60 subjects
Exploratory: For each vaccine group the antibody responses to the H5 vaccine strain evaluated by single radial hemolysis (SRH) assay | Days 0 and 63 (21 days after the H5N1 immunization)
  All subjects
Exploratory: The association between cellular immune markers and humoral immune responses will be examined. | Days 0, 42 and 63

CONTACTS AND LOCATIONS:
Overall Officials: Dora Mathiasz, MD, Study Director — St Istvan St Laszlo hospital
Locations (1):
- St Istvan St laszlo Hospital, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
summary of data per group will be shared, not IPD.